CLINICAL TRIAL: NCT07117032
Title: A Prospective Pilot Clinical Trial of Simulation-Free Celiac Plexus Pain Ablation Using Stereotactic Body Radiotherapy in Patients With Cancer-Related Celiac Pain
Brief Title: Simulation-Free Celiac Plexus Pain Ablation Using Stereotactic Body Radiotherapy (SBRT) in Participants With Cancer-Related Celiac Pain
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE5225
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Pancreatic Cancer; Retroperitoneal Pain Syndrome
Keywords: Abdominal pain; Stereotactic Body Radiotherapy; Celiac pain; Celiac plexus pain ablation; SBRT
MeSH Terms: conditions — Pancreatic Neoplasms; Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Simulation-free treatment delivery of celiac plexus SBRT (Experimental)
  Interventions: Other: Simulation-free workflow; Radiation: Celiac plexus SBRT

INTERVENTIONS:
Other: Simulation-free workflow — Pre-existing diagnostic images (CTs, PET/CTs, or MRIs) will be imported into the online treatment planning system called Ethos. The Ethos platform and online adaptive radiation therapy (ART) will be utilized at the time of treatment planning and delivery.
Radiation: Celiac plexus SBRT — Participants will receive SBRT per standard of care. This treatment visit will take up to 1.5 hours.

SUMMARY:
Participants who are experiencing abdominal pain due to having cancer in their pancreas may be eligible for this research study. For this type of pain, doctors often recommend radiation therapy to help with the pain. This radiation therapy is called stereotactic body radiotherapy (SBRT). Preparing for SBRT typically takes a week or longer. In this research study, doctors want to test a new workflow in order to shorten the time it takes for participants to receive SBRT to help with their pain.

Doctors typically determine how to administer the SBRT by doing a simulation, which requires a CT (Computerized Tomography) scan. The CT scan is used to create a treatment plan. It can take time to schedule this CT scan and then it takes 5-10 days to create a treatment plan. A way to reduce the planning time for SBRT is to use the CT scan that participants had when their cancer was diagnosed to plan the SBRT. This new workflow can cut down the time it takes to schedule another CT scan and plan for and deliver SBRT. The workflow where doctors use a pre-existing CT scan is called CTsim-free treatment planning. CTsim-free treatment planning is what is being tested in this research study.

DETAILED DESCRIPTION:
Celiac plexus nerve pain, a type of abdominal pain, is common in people with pancreatic cancer. In fact, 70-80% of these people say they have very bad, or debilitating, pain in the lower part of their abdomen and/or the area behind their abdomen where they were diagnosed with pancreatic cancer (1). Recently, a type of treatment called celiac plexus radioablation, which is done using a type of radiation called stereotactic body radiotherapy (SBRT), has been recognized as a new standard-of-care therapy option for these people (2-4).

However, celiac plexus radioablation takes a long time to plan and deliver when compared to traditional treatment approaches, which don't require so much time and so many visits (5). A better workflow is needed to make treatment planning and delivery happen faster. This better workflow should make things easier on people who are experiencing this severe pain and help them start treatment faster to feel better sooner.

One way to create this better workflow for celiac plexus radioablation is to use single-fraction SBRT and to use simulation-free radiation treatment planning. For this type of workflow, pre-existing diagnostic images are used to make the treatment plan, rather than making people get new images before they can start getting treated for their pain (6). This workflow uses an online tool called online adaptive radiotherapy (ART) to help create and adjust the treatment plan based on what can be seen inside the body on the pre-existing diagnostic images so that it targets the right spot.

The research study team has developed an institutional celiac plexus auto-planning template using a commercial CT-guided ART platform. The team has looked back at past cases and confirmed that this workflow can safely create treatment plans in a short amount of time. The adaptive radiotherapy that is used in this simulation-free workflow is a a standard-of-care practice for other disease sites. There have been previous research studies that show that it works to lessen the time to treatment when treating other areas of the body (7-9).

The novel approach in this study is the workflow, and as such, the purpose of this study is to demonstrate the feasibility and safety of a simulation-free workflow for celiac plexus SBRT using online adaptive radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed cancer that is metastatic or unresectable, and considered appropriate per the treating physician to receive celiac plexus SBRT.
* Age >18 years. Because no data are currently available on the use of celiac axis SBRT in participants ≤18 years of age, children are excluded from this study.
* Performance status: ECOG Performance status ≤ 3
* Severe retroperitoneal pain syndrome (radiates from the lower back to the upper abdomen, belt- like distribution), intensity of at least 5 on 11-point Brief Pain Inventory (BPI, average pain) scale despite analgesic use. Note: previous use of celiac plexus block/neurolysis for pain control is allowed and will be recorded
* Participants must have anatomical involvement of the celiac plexus on the diagnostic CT, PET/CT, or MRI. This includes:

  * Any pancreatic cancer
  * Any other cancer that on imaging demonstrates either gross involvement of the celiac blood vessels or celiac plexus on imaging OR haziness around the celiac blood vessels that typically implies tumor engulfment.
* Prior chemotherapy or biological treatment is allowed, but any active oncological treatment must be stopped at least 1 week prior to radiation therapy and renewed at least 1 week following radiation therapy.
* Participants must have the ability to understand and the willingness to sign a written informed consent document.
* Participants must have a diagnostic CT, PET/CT, or MRI of the abdomen and pelvis, with or without contrast, acquired < 28 days prior to the study consent. This diagnostic scan, to be used for pre-plan formation, must fully visualize the celiac plexus target intended for simulation-free treatment, with full axial field-of-view at the axial levels for treatment. The scan must be of sufficient clinical quality for the treating physician to delineate the target for treatment.

Exclusion Criteria:

* Prior radiotherapy to the upper abdomen.
* Previous radiotherapy to the upper abdomen overlapping with the projected site of treatment.
* Pregnant or breastfeeding women are excluded from this study.
* Participants with conditions associated with increased risk of side effects from radiation such as inflammatory bowel disease and scleroderma.
* Women of childbearing potential must have a negative pregnancy test within 14 days of study entry. If pregnancy test is not clinically indicated as determined by treating physician or protocol principal investigator, documentation of this exception is sufficient in lieu of a pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the simulation-free adaptive radiotherapy workflow, as measured by rate of successful completion of treatment | At treatment visit, 1.5 hours
  Successful completion is defined as completion of the simulation-free ART workflow through treatment delivery in the first on-table treatment attempt for at least 80% of participants with simulation-free plans meeting dosimetric requirements.
Feasibility of the simulation-free adaptive radiotherapy workflow, as measured by rate of compliance with priority level 1 dose constraints | At treatment visit, 1.5 hours
  Compliance with priority level 1 dose constraints is defined as having a pre-treatment quality assurance clinical gamma passing index less than or equal to 2%/ 2mm.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Henke, MD, MSCI, Principal Investigator — Case Comprehensive Cancer Center, University Hospitals
Locations (1):
- University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Molnar I, Hegyi G, Zsom L, Saahs C, Vagedes J, Kapocs G, Kovacs Z, Sterner MG, Szoke H. Celiac plexus block increases quality of life in patients with pancreatic cancer. J Pain Res. 2019 Jan 14;12:307-315. doi: 10.2147/JPR.S186659. eCollection 2019. PMID 30679920
- [Background] Hammer L, Hausner D, Ben-Ayun M, Shacham-Shmueli E, Morag O, Margalit O, Boursi B, Yarom N, Jacobson G, Katzman T, Abrams R, Dicker A, Golan T, Symon Z, Lawrence YR. Single-Fraction Celiac Plexus Radiosurgery: A Preliminary Proof-of-Concept Phase 2 Clinical Trial. Int J Radiat Oncol Biol Phys. 2022 Jul 1;113(3):588-593. doi: 10.1016/j.ijrobp.2022.02.038. Epub 2022 Mar 4. PMID 35257800
- [Background] Jacobson G, Fluss R, Dany-BenShushan A, Golan T, Meron T, Zimmermann C, Dawson LA, Barry A, Miszczyk M, Buckstein M, Diaz Pardo D, Aguiar A, Hammer L, Dicker AP, Ben-Ailan M, Morag O, Hausner D, Symon Z, Lawrence YR. Coeliac plexus radiosurgery for pain management in patients with advanced cancer : study protocol for a phase II clinical trial. BMJ Open. 2022 Mar 24;12(3):e050169. doi: 10.1136/bmjopen-2021-050169. PMID 35332036
- [Background] Lawrence YR, Miszczyk M, Barry AS, Diaz Pardo DA, Aguiar A, Limon D, et al. Celiac plexus radiosurgery for pain management in advanced cancer: An international phase II trial, health-related quality of life (HRQOL) outcomes. American Society of Clinical Oncology; 2023.
- [Background] Lo SS, Fakiris AJ, Chang EL, Mayr NA, Wang JZ, Papiez L, Teh BS, McGarry RC, Cardenes HR, Timmerman RD. Stereotactic body radiation therapy: a novel treatment modality. Nat Rev Clin Oncol. 2010 Jan;7(1):44-54. doi: 10.1038/nrclinonc.2009.188. Epub 2009 Dec 8. PMID 19997074
- [Background] Schuler T, Back M, Hruby G, Carroll S, Jayamanne D, Kneebone A, Stevens M, Lamoury G, Morgia M, Wong S, Grimberg K, Roderick S, Booth J, Eade T. Introducing Computed Tomography Simulation-Free and Electronic Patient-Reported Outcomes-Monitored Palliative Radiation Therapy into Routine Care: Clinical Outcomes and Implementation Experience. Adv Radiat Oncol. 2020 Dec 3;6(2):100632. doi: 10.1016/j.adro.2020.100632. eCollection 2021 Mar-Apr. PMID 33851063
- [Background] Wong S, Roderick S, Kejda A, Atyeo J, Grimberg K, Porter B, Booth J, Hruby G, Eade T. Diagnostic Computed Tomography Enabled Planning for Palliative Radiation Therapy: Removing the Need for a Planning Computed Tomography Scan. Pract Radiat Oncol. 2021 Mar-Apr;11(2):e146-e153. doi: 10.1016/j.prro.2020.10.010. Epub 2020 Nov 10. PMID 33186781
- [Background] Schiff JP, Zhao T, Huang Y, Sun B, Hugo GD, Spraker MB, Abraham CD. Simulation-Free Radiation Therapy: An Emerging Form of Treatment Planning to Expedite Plan Generation for Patients Receiving Palliative Radiation Therapy. Adv Radiat Oncol. 2022 Oct 3;8(1):101091. doi: 10.1016/j.adro.2022.101091. eCollection 2023 Jan-Feb. PMID 36304132
- [Background] Nelissen KJ, Versteijne E, Senan S, Rijksen B, Admiraal M, Visser J, Barink S, de la Fuente AL, Hoffmans D, Slotman BJ, Verbakel WFAR. Same-day adaptive palliative radiotherapy without prior CT simulation: Early outcomes in the FAST-METS study. Radiother Oncol. 2023 May;182:109538. doi: 10.1016/j.radonc.2023.109538. Epub 2023 Feb 16. PMID 36806603